CLINICAL TRIAL: NCT06105723
Title: An Effectiveness Evaluation for Pathway to Healthy Aging (Path-HA) Care on Health Status of Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Yu, Doris Sau Fung, Professor (Chair, Research), The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PATHHA
Record Dates: First submitted 2023-10-23; First posted 2023-10-30 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Ageing Well
Keywords: Aging; Functional ability; Care model; Community-dwelling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Path-HA care (Experimental): A 14-week care initiative comprising two phases is provided, which are the 2-week ICOPE-based personalized care planning phase, and the 12-week healthy aging empowerment phase.
  Interventions: Behavioral: Pathway to Healthy Aging care
- Control (No Intervention): No care intervention will be provided.

INTERVENTIONS:
Behavioral: Pathway to Healthy Aging care — The ICOPE-based personalized care planning comprises two home visits. In 1st visit, a comprehensive assessment proposed by the WHO-ICOPE model is conducted to identify eight possible health problems including malnutrition, reduced physical fitness, fall risk, cognitive decline, insomnia, pain, psychological distress and social loneliness. After health problem identification, each participant receives a personalized care prescription. 2nd visit adopts a goal-oriented empowerment 3-step cycle to personalize the care planning: 1) communicating assessment results to increase healthy self-awareness; 2) supporting setting person-directed goals to address health problems; 3) identifying health actions and personalizing goal setting to participants' contexts. The 12-week healthy aging empowerment comprises three core activities for healthy aging promotion, including interactive health education, health message broadcasts, and three case conferences for goal monitoring and health counseling.
  Arms: Path-HA care

SUMMARY:
The goal of this clinical trial is to provide a scientific evaluation on the effects of a protocol-driven Pathway to Healthy Aging (Path-HA) Program on promoting the health-related quality of life and functional abilities of older adults who are at risk of accelerated aging in the community. Participants will be randomized to one of the two study arms: 1) the intervention group to receive a 14-week Path-HA care intervention; and 2) the control group with no Path-HA care intervention.

DETAILED DESCRIPTION:
This assessor-blind, randomized controlled trial evaluates the effects of the Pathway to Healthy Aging Program, which is based on the WHO ICOPE model, on the promotion of the health-related quality of life (primary outcome) as well as functional abilities (secondary outcomes) as defined by the WHO-ICOPE among community-dwelling older adults with accelerated aging. Six health domains including locomotor function, vitality, psychological function, cognitive function, social functions, and overall health-related quality of life are measured. A total of 1000 participants will be recruited. Outcome evaluation takes place at baseline, upon the completion of the care program, and at 6 months thereafter to allow the detection of long-term program benefits. In-depth individual interviews will be conducted to solicit the participants' experience and perceived benefits of the program.

ELIGIBILITY:
Inclusion Criteria:

* 1) aged 60 or above,
* 2) with at least two risk factors of accelerating aging defined as including reduced physical functioning, malnutrition, depressed mood, loneliness, poor health perception, and presence of geriatric symptoms (e.g. insomnia, pain, etc), based on their health screening results,
* 3) community-dwelling,
* 4) communicable to engage in health education activity.

Exclusion Criteria:

* 1) any who is not at or at only one risk factor of accelerating aging,
* 2) any who has problems in communicating with the research team.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life | Changes from baseline to 3-month and 9-month post-intervention
  Measured by the EQ-5D-5L questionnaire (scores range from -0.59 to 1.0), with a higher score indicating better quality of life.

SECONDARY OUTCOMES:
Hand grip strength | Changes from baseline to 3-month and 9-month post-intervention
  Measured by hand-held dynamometer in unit of KG. A larger count indicates a greater grip strength.
Balancing function | Changes from baseline to 3-month and 9-month post-intervention
  Measured by the Timed Up and Go Test in unit of second. A shorter completion time indicates better mobility and balance.
Physical mobility level | Changes from baseline to 3-month and 9-month post-intervention
  Measured by the Short Physical Performance Battery (scores range from 0 to 12), with higher scores indicating better physical performance and better mobility functioning.
Sarcopenia risk | Changes from baseline to 3-month and 9-month post-intervention
  Measured by Sarcopenia and calf circumference scale (SARC-CalF scale). The score ranges from 0 to 20 points, with a score ≥ 11 points suggestive of sarcopenia.
Nutritional status | Changes from baseline to 3-month and 9-month post-intervention
  Measured by the Mini Nutritional Assessment (scores range from 0 to 30), with a lower score indicating a higher risk of malnutrition.
Sleep quality | Changes from baseline to 3-month and 9-month post-intervention
  Measured by Insomnia Severity Index questionnaire (scores range from 0 to 28), with higher scores indicating greater severity of insomnia.
Depressed mood | Changes from baseline to 3-month and 9-month post-intervention
  Measured by the 15-item Geriatric Depression Scale (scores range from 0 to 15), with a higher score indicating a higher risk of depression.
Cognitive functions | Changes from baseline to 3-month and 9-month post-intervention
  Measured by the 5-minute Montreal Cognitive Assessment Test (scores range from 0 to 30). A raw score of < 25 in well-educated persons (education > 12 years) or a raw score of < 23 in less-educated persons (education ≤ 12 years) is defined as impaired cognition.
Subjective memory | Changes from baseline to 3-month and 9-month post-intervention
  Measured by Memory Inventory for the Chinese (scores range from 0 to 108), with higher scores indicating more severe subjective memory loss.
Loneliness | Changes from baseline to 3-month and 9-month post-intervention
  Measured by The 3-Item UCLA Loneliness Scale (scores range from 3 to 9), with higher scores suggesting a higher level of loneliness.
Social connectedness | Changes from baseline to 3-month and 9-month post-intervention
  Measured by The 8-item version of Social Connectedness Scale (scores range from 8 to 48), with a higher score indicating a greater sense of social connectedness.

CONTACTS AND LOCATIONS:
Overall Officials: Doris Sau Fung YU, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong